CLINICAL TRIAL: NCT07319637
Title: Comparison of the Outcome of Orchidopexy With and Without Sac Ligation in Paediatric Population With Palpable Undescended Testis
Brief Title: Comparing Two Types of Surgery for Children With Undescended Testicles When the Hernia Sac Is Tied or Not
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children Hospital Faisalabad (Other)
Responsible Party: Principal Investigator, Rida Dawood, Postgraduate Resident, Children Hospital Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPSP/REU/PSG-2023-290-572; No.32/CH&ICH/FSD, 16-Jan-2024 (Other: Children Hospital & Institute of Child Health, Faisalabad.)
Record Dates: First submitted 2025-12-09; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Undescended Testis
Keywords: Orchiopexy; sac ligation; Palpable Undescended testis
MeSH Terms: conditions — Cryptorchidism | interventions — Orchiopexy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Orchiopexy with sac ligation
  Interventions: Procedure: Orchiopexy with sac ligation
- Group B (Experimental): Orchiopexy without sac ligation
  Interventions: Procedure: Orchiopexy without sac ligation

INTERVENTIONS:
Procedure: Orchiopexy without sac ligation — To compare the outcome of the surgery with and without sac ligation in pediatric population with palpable undescended testes.
  Arms: Group B
Procedure: Orchiopexy with sac ligation — To compare the outcome of the surgery with and without sac ligation in pediatric population with palpable undescended testes.
  Arms: Group A

SUMMARY:
When a child has an undescended testicle that can be felt in the groin, surgery (orchiopexy) is needed to move it into the scrotum. During this operation, doctors sometimes tie off a small sac near the testicle, but this step can make the surgery longer and may slightly increase risks like swelling, infection, or irritation.

This study looks at whether tying this sac is really necessary. It compares children who had surgery with sac ligation to those who had surgery without it. The goal is to see if there is any difference in surgery time or the chance of developing a hernia afterward. By understanding this, doctors can choose the safest and simplest approach for children with undescended testicles and provide better care.

DETAILED DESCRIPTION:
Cryptorchidism or Undescended testis (UDT) is described as testes that cannot be brought down to the bottom of scrotum without undue traction on the spermatic cord. It is one of the most common conditions presenting in pediatric surgical outpatient department1. UDT is seen in 2-4% of children at birth, decreasing to about 1% in the first year of life. It is prevalent in about one to four and a half percentage of newborns with a higher incidence in preterm babies (30-45%). UDT maybe unilateral or bilateral, mostly affecting the right side (70%).

The management of palpable undescended testes (UDT) in the pediatric population often necessitates surgical intervention to relocate the testes into the scrotum, a procedure known as orchiopexy. During this surgery, surgeons may choose to either ligate the hernia sac associated with the undescended testis or leave it unligated. The decision to ligate the sac is influenced by the belief that it might reduce the risk of post-operative complications such as inguinal hernias. However, this additional step could potentially prolong the operative time and introduce other risks.

Studies suggest there is probability of spontaneous decent in the first three months postnatally, beyond which it was rare. The recommended age for surgery for undescended testis is six months of age. The standard surgical intervention for orchiopexy was described in 1881-1899. The classical orchidopexy recommends the mandatory ligation of the hernial sac to prevent occurrence of postoperative hernia. This traditional conventional orchidopexy technique is well-acknowledged and generally practiced and is well supported by many studies that conclude that sac ligation is mandatory for the prevention of post-operative complication of inguinal hernia5. However, recent evidence advocates that orchidopexy with ligation of hernial sac is unnecessary procedure with increased occurrence of severe pain post-operatively along with increased chances of testicular atrophy due to inadvertent injury to the adjacent structures6. Furthermore, it has been found that orchidopexies without ligation of sac technique is simple, save intraoperative time and equally effective with comparable outcomes.

A recent study on orchidopexy with and without sac ligation in pediatric patients was conducted to compare mean operative time and incidence of complications including post-operative hernia A total of hundred patients were recruited in this study. In one group orchidopexy without dissection and ligation of peritoneal sac was done, while in other group included the patients in which sac ligation was performed. In this study 60 (60%) patients had left-sided whereas 40 (40%) patients had right-sided UDT. The mean operative time of the patients from no sac ligation group was 21.25±0.90 minutes whereas in ligation group 33.10±1.10 minutes. Interestingly, no case of post-operative hernia was noted in both groups (0.00%).

Rationales of the study: The surgical management of palpable undescended testes (UDT) in children involves the critical decision of whether to ligate the associated hernia sac, a step that may prolong operative time and introduce additional risks such as inflammation, infection, or tissue damage. This study aims to evaluate the impact of sac ligation on operative time and the incidence of post-operative inguinal hernias, providing a comprehensive risk-benefit analysis. By comparing the outcomes of pediatric orchiopexy with and without sac ligation, the study seeks to generate high-quality evidence to guide surgical practice, standardize care, and ultimately improve patient outcomes and healthcare resource utilization in the treatment of palpable UDT.

OBJECTIVES: To compare the outcome (in terms of operative time and occurrence of post operative inguinal hernia) of the surgery with and without sac ligation in pediatric population with palpable undescended testes.

ELIGIBILITY:
Inclusion Criteria:

* Male children ≤15 years with palpable UDT
* Scheduled for single stage orchidopexy

Exclusion Criteria:

* Impalpable testes
* Staged/laparoscopic procedures,
* Pre-op hernia,
* History previous orchiopexy
* Ambiguous genitalia

Ages: 6 Months to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Operative Time | During surgery "from skin incision to skin closure", assessed at the time of the surgical procedure.
Post-operative Complications | at 0, 4, 8 and 12 weeks after surgery
  Post-op hernia, Wound infection, Hematoma and Testicular atrophy

SECONDARY OUTCOMES:
Hospital stay duration, or Length of Stay (LOS) in the hospital | From the day of the admission for procedure until hospital discharge, assessed during the index hospitalization (up to 7 days)
Post-operative Pain Score | Post-operative period, assessed at 3 hours, 6 hours, 12 hours, 24 hours, and 48 hours after surgery.
  Pain intensity will be assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores represent greater pain severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital & Institute of Child Health, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No